CLINICAL TRIAL: NCT05347173
Title: Dexmedetomidine Versus Nalbuphine as an Adjuvant to Intrathecal Bupivacaine in Lower Limb Surgeries
Brief Title: Dexmedetomidine Versus Nalbuphine as an Adjuvant to Intrathecal Bupivacaine
Acronym: Intrathecal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Assistant Professor of Anesthesia and Surgical Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dexmed+Nalbuph
Record Dates: First submitted 2022-04-13; First posted 2022-04-26 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Nalbuphine

STUDY DESIGN:
Intervention Model Description: Via the sealed envelope method; the patients will be randomly assigned to three equal groups according to the administration of adjuvant to intrathecal Bupivacaine and its dose;
  * Bupivacaine group (B gp) will include patients who will receive 2.5 ml hyperbaric bupivacaine (0.5%) +0.5 ml normal saline.
  * Bupivacaine-Dexmedetomidine group (BDgp) will include patients who will receive 2.5 ml hyperbaric bupivacaine (0.5%) plus Dexmedetomidine (10 µg in 0.5 ml normal saline).
  * Bupivacaine-Nalbuphine group (BN gp) will include patients who will receive 2.5 ml hyperbaric bupivacaine (0.5%) plus Nalbuphine (1 mg in 0.5ml normal saline).
Who Masked: Participant, Investigator
Masking Description: Intrathecal injectate will be prepared according to the group by an anesthesiologist who is not involved in data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bupivacaine group (B gp) (No Intervention): Patients will receive 2.5 ml hyperbaric bupivacaine (0.5%) plus 0.5 ml normal saline
- Bupivacaine-Dexmedetomidine group (BD gp) (Active Comparator): Patients will receive 2.5 mL hyperbaric bupivacaine (0.5%) plus 10 µg Dexmedetomidine in 0.5 mL normal saline
  Interventions: Drug: Dexmedetomidine
- Bupivacaine-Nalbuphine group (BN gp) (Active Comparator): Patients will receive 2.5 mL hyperbaric bupivacaine (0.5%) plus 1 mg Nalbuphine in 0.5 mL normal saline
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: Dexmedetomidine — patients who will receive 2.5 mL hyperbaric bupivacaine (0.5%) plus Dexmedetomidine (10 µg in 0.5 mL normal saline)
  Arms: Bupivacaine-Dexmedetomidine group (BD gp)
Drug: Nalbuphine — patients who will receive 2.5 mL hyperbaric bupivacaine (0.5%) plus Nalbuphine (1 mg in 0.5 mL normal saline)
  Arms: Bupivacaine-Nalbuphine group (BN gp)

SUMMARY:
Spinal anesthesia is the most consistent block for lower abdomen and lower limb surgical procedures. Over years many drugs have been used as an additive to spinal anesthesia in order to prolong the duration of action and to provide adequate postoperative analgesia.

Dexmedetomidine, a highly selective α2 agonist is rapidly emerging as the choice of additive to spinal anesthesia in view of its property to provide analgesia however, it may be associated with bradycardia which may affect the hemodynamic stability.

Nalbuphine is an opioid with agonist actions in the kappa receptor and antagonist actions in the mu receptor, it produces analgesia and sedation and lesser side effects through antagonism at the mu receptor but, it could be associated with some side effects as: dizziness, bradycardia, nausea, vomiting, and pruritus and may be associated with respiratory depression.

DETAILED DESCRIPTION:
This prospective, double blinded, randomized, controlled study will be held to compare Nalbuphine versus Dexmedetomidine as adjuvants to intrathecal Bupivacaine in spinal anesthesia in patients undergoing lower limb orthopedic surgeries

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60 years.
* Both genders.
* Patients scheduled for lower limb orthopedic surgeries under spinal anesthesia.
* American society of anesthesiologists (ASA) class I or II.

Exclusion Criteria:

* Patient refusal.
* Age <20 or >60 years.
* Contraindications to spinal anesthesia (e.g. bleeding diathesis, spinal cord deformities, infection at injection site).
* History of allergy to any of the study medications.
* Cases with severe cardiac, renal, or hepatic disease.
* American society of anesthesiologists (ASA) class III, IV.
* Patient on regular analgesics or opioid abuse.
* Patient with peripheral neuropathy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
The post-operative analgesic duration | during the first 24 postoperative hours

SECONDARY OUTCOMES:
Onset of sensory block | After intrathecal injection up to 15 minutes
  from intrathecal injection till sensory block grade 2 at T10
Onset of motor block | After intrathecal injection up to 15 minutes
  from intrathecal injection till reach Bromage scale 3
Heart rate (HR) | Every 5 minutes after spinal injection for the first 30 minutes, and then every 15 minutes till the end of surgery
  beat per minute
Mean arterial pressure (MAP) | Every 5 minutes after spinal injection for the first 30 minutes, and then every 15 minutes till the end of surgery
  mmHg
Hypotension will be considered if there was 25% decrease below the baseline for Mean arterial pressure (MAP) | every 5 minutes after spinal injection for the first 30 minutes, then every 15 minutes till the end of surgery and every 30 minutes for the first 6 hours postoperatively
  mmHg
Bradycardia will be considered if the heart rate is less than 50 beats/min | every 5 minutes after spinal injection for the first 30 minutes, then every 15 minutes till the end of surgery and every 30 minutes for the first 6 hours postoperatively
  beat per minute
postoperative pain | at 0, 2, 4, 6, 8,12,18 and 24 hours postoperatively
  visual analogue scale (VAS) marked from 0-10 (where 0 = no pain and 10 = worst pain imaginable)
side effects as Vomiting, Nausea, pruritus, shivering | Intraoperatively and for the first 24 hours postoperatively
  incidence
sedation | at 0, 2, 4, 6, 8,12,18 and 24 hours postoperatively
  via Ramsay scale [1= Patient is anxious and agitated or restless, or both, 2= Patient is co-operative, oriented, and tranquil, 3= Patient responds to commands only, 4= Patient exhibits brisk response to light glabellar tap or loud auditory stimulus, 5= Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus and 6=Patient exhibits no response]

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University-Emergency hospital-ICU, El Dakahlia, Mansoura, Egypt